CLINICAL TRIAL: NCT05871242
Title: Study to Investigate the Treatment Benefit of Probiotic Lactobacillus Crispatus M247 in Women Undergoing Homologous Level 2 Assisted Reproductive Technology (ART) Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Amjad Khan (Other)
Collaborators: Treviso Regional Hospital (Network)
Responsible Party: Sponsor-Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Organization: Liaquat University of Medical & Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUMHS/REC/-253
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Fertility Issues
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Treatment with Lactobacillus crispatus M247
  Interventions: Dietary Supplement: Probiotic Lactobacillus crispatus M247
- Control arm (No Intervention): No Probiotic treatment

INTERVENTIONS:
Dietary Supplement: Probiotic Lactobacillus crispatus M247 — Patient who have received probiotic Lactobacillus crispatus M247
  Arms: Treatment arm

SUMMARY:
The present study is aimed to explore the treatment effect from the intake of probiotic Lactobacillus crispatus M247 in the improvement of clinical and psychological aspects in women undergoing homologous level 2 ART procedures.

DETAILED DESCRIPTION:
The use of assisted reproductive technology (ART) has increased dramatically worldwide due to the continuous rise in infertility rates; for these reasons an increasing number of couples undertake the path of ART, even though this is difficult journey, with uncertain outcomes and possible medical risks, both physical and psychological.

In this study the investigators aim to explore the hypothesis that recreating a favorable vaginotype through the intake of the probiotic Lactobacillus crispatus M247 can have a positive effect in achieving pregnancy in cryopreserved cycles as well as a positive relationship between vaginal, endometrial (still unknown), gut and oral microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing homologous level 2 assisted reproductive technology (ART) procedures
* Cryopreserved oocytes
* D3 embryos
* D5 blastulae
* Age 18-45

Exclusion Criteria:

* Presence of submucous uterine myomas.
* Uterine malformations.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study is applicable only to women
Enrollment: 160 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy | up to 12 months
  Rate of pregnancy

SECONDARY OUTCOMES:
Effect on sex hormonal profile | up to 12 months
  change in anti-mullerian hormone levels
Effect on sex hormonal profile | up to 12 months
  Change in Follicle Stimulating Hormone levels
Effect on sex hormonal profile | up to 12 months
  Change in Free testosterone levels

CONTACTS AND LOCATIONS:
Locations (1):
- ART center, Hospital of Conegliano, Treviso, Italy